CLINICAL TRIAL: NCT02202109
Title: Addressing Cervical Cancer Disparity in South Florida: CBPR in Action
Brief Title: Using CHWs or Mailing Self Sampling Home Tests to Increase Cervical Cancer Screening in South Florida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Health Choice Network (Other); Center for Haitian Studies (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erin Kobetz-Kerman, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20140249; 1R01CA183612-01 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-28 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cervical Cancer
Keywords: Screen; self-sampler; cervical, cancer; women; community health workers; Hispanic/ Latinas; Haitian; Focus of study is cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHWs facilitated Self-Sampling (Active Comparator): CHW and Self-sampling for Cervical Cancer. Home visit, self-sampler, collection of test
  Interventions: Behavioral: CHW and Self-sampling for Cervical Cancer
- Mailed Self-Sampler (Active Comparator): Mailed Self Sampler. Self sampler is mailed to participant; follow up by phone
  Interventions: Behavioral: Mailed Self Sampler

INTERVENTIONS:
Behavioral: CHW and Self-sampling for Cervical Cancer — Behavioral: CHW and Self-sampling for Cervical Cancer The intervention strategies will involve one home visit: 1) provide brief health education on cervical cancer screening, 2) provide and collect self-sampler test. We envision visits lasting no more than 60 minutes.
  Arms: CHWs facilitated Self-Sampling
Behavioral: Mailed Self Sampler — Mailed Self Sampler. Women randomized to this intervention arm will receive a self-sampling kit via mail. This kit will include: 1) the self-sampler; 2) the vial for collecting and storing the specimen; 3) a pre-addressed, stamped envelope for returning the vial; 4) a brief introductory letter/postcard which includes a picture of the CHE and the CHW and serves to re-orient the participant to the focus of the study; 5) instructional guide that visually depicts the steps for self-sampling;
  Arms: Mailed Self-Sampler

SUMMARY:
The study will test the significance of community health worker (CHW) participation by comparing self-sampling provided by a community health worker and self-sampling provided by mail. The study will enroll 700 participants in communities that lack access to medical care in South Florida.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Haitian, Hispanic, or African American
* Ages 30-65 years
* Report not having had a pap smear in the last three years live in the cities of Miami/Little Haiti, Hialeah or unincorporated Southern Miami-Dade

Exclusion Criteria:

* Women who report having had a hysterectomy
* Women who have a history of cervical cancer
* Women who plan to move outside of Miami-Dade county during the next six months
* Women who are enrolled in any other cancer prevention/outreach related study
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Kobetz, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Kobetz E, Seay J, Amofah A, Pierre L, Bispo JB, Trevil D, Gonzalez M, Poitevien M, Koru-Sengul T, Carrasquillo O. Mailed HPV self-sampling for cervical cancer screening among underserved minority women: study protocol for a randomized controlled trial. Trials. 2017 Jan 13;18(1):19. doi: 10.1186/s13063-016-1721-6. PMID 28086983

RESULTS

PARTICIPANT FLOW:
Groups:
- CHWs Facilited Self-Sampling: CHW and Self-sampling for Cervical Cancer. Home visit, self-sampler, collection of test
  CHW and Self-sampling for Cervical Cancer: Behavioral: CHW and Self-sampling for Cervical Cancer The intervention strategies will involve one home visit: 1) provide brief health education on cervical cancer screening, 2) provide and collect self-sampler test. We envision visits lasting no more than 60 minutes.
Period: Overall Study
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler
Started | 302 | 300
Completed | 212 | 213
Not Completed | 90 | 87
Not completed — Lost to Follow-up | 88 | 87
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler | Total
Number analyzed (Participants) | 302 | 300 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 302 | 300 | 602
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 300 | 602
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 198 | 197 | 395
  Not Hispanic or Latino | 103 | 103 | 206
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 106 | 113 | 219
  White | 141 | 138 | 279
  More than one race | 54 | 47 | 101
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing a Self-sampling Test
Description: The primary outcome is having had a self-sampling done since the initial evaluation. Participants who test negative will be encouraged to rescreen while Participants who test positive for HPV will be navigated to appropriate follow-up care. The CHWs will follow up with participants who do not return the kit within 60 days.
Time Frame: 2 to 6 months
Population: Participants were given up to 6 months to complete HPV self-sampling.
Measure: Count of Participants; unit: Participants
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler
Number analyzed (Participants) | 272 | 257
Participants | 272 | 257

2. Secondary Outcome: Proportion of Change in Cervical Cancer Knowledge Among Participants
Description: Cervical cancer knowledge was measured with a series of questions asked at both pre(baseline) and post (exit). The questions were designed to measure participant's knowledge of cervical cancer prior to the study intervention and following the intervention. Cervical cancer knowledge is defined by participants answering 3 out 5 questions correctly.
Time Frame: Baseline, 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler
Number analyzed (Participants) | 212 | 213
proportion of participants | 0.033 [-0.038 to 0.104] | 0.089 [0.017 to 0.162]

3. Secondary Outcome: Proportion of Participants With a Change in Access to Care
Description: Access to care was defined as having a routine source of care and measured at both pre(baseline) and post (exit).
Time Frame: Baseline, 6 months
Population: Only participants with complete information on access to care were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler
Number analyzed (Participants) | 212 | 211
proportion of participants | 0.160 [0.092 to 0.230] | 0.166 [0.088 to 0.244]

ADVERSE EVENTS:
Time Frame: Data for adverse events was collected for a period of one year.
Arm/Group | CHWs Facilited Self-Sampling | Mailed Self-Sampler
All-Cause Mortality (participants affected / at risk) | 0/302 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/302 | 0/300
Other Adverse Events (participants affected / at risk) | 0/302 | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT02202109/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02202109/SAP_001.pdf